CLINICAL TRIAL: NCT06702371
Title: EMBody ('Exploring Mindsets About the Body'): Harnessing Adaptive Body Mindsets to Improve Outcomes in Childhood & AYA Cancer Survivors
Brief Title: Digital Body Mindset Intervention for Young Cancer Survivors
Acronym: EMBody
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 324319; MRF-015-0001-RG-HEAT-C0955 (Other Grant/Funding Number: Medical Research Foundation)
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Childhood Cancer; Survivors of Childhood Cancer; Mindsets; Mindset Intervention; Adolescent and Young Adult (AYA); Wise Intervention; Body Mindsets
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated (1:1) to the EMBody intervention group or the waitlist attention control group. Those in the intervention group will complete the EMBody intervention content as well as online surveys. Those in the control group will complete the online surveys at the same time points and will receive the EMBody intervention content after their study involvement.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocation concealment is ensured through the use of Sealed Envelope, which maintains the randomisation schedule securely and prevents members of the research team responsible for enrolling participants from accessing the allocation sequence. The research team involved in data collection will not be blinded to group allocation. Members of the research team who will analyse the data will be blinded to the randomisation schedule and group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindset Intervention (Experimental): Participants who are randomised to the intervention arm will complete all three modules of the EMBody intervention across six weeks. They will also complete online surveys at baseline (T0), weeks two (T1), four (T2), six (T3), 10 (T4), and 18 (T5). Data will be analysed after the T5 data collection point. There will be an additional 12-month long-term follow up (T6), with a go/no-go decision depending on trial findings; these data will be published separately.
  Interventions: Behavioral: Mindset Intervention
- Waitlist Attention Control (No Intervention): Participants randomised to the waitlist attention control arm will complete the online surveys at the same timepoints as participants randomised to the intervention arm. After the 12-month long-term follow-up survey (T6), participants in the waitlist control arm will be sent the EMBody intervention materials.

INTERVENTIONS:
Behavioral: Mindset Intervention — The EMBody intervention contains seven short documentary-style films and paired reflection activities across three modules.
  Module 1: Introducing Mindsets (Film 1: A New normal; Film 2: What is a Mindset?; Film 3: Your Body is Capable; Film 4: How to Choose Your Mindset).
  Module 2: Challenges and Setbacks (Film 5: Living with Uncertainty; Film 6: The Long and Winding Road).
  Module 3: Looking to the Future (Film 7: Opportunities Emerge).
  Arms: Mindset Intervention

SUMMARY:
The aim of this study is to assess whether a digital body mindset intervention - EMBody - can instil adaptive mindsets and improve health and wellbeing in young cancer survivors aged 16-25.

DETAILED DESCRIPTION:
EMBody (Exploring Mindsets about the Body) is a brief digital intervention comprising documentary-style films and reflection activities which aim to instil adaptive mindsets in young people who have previously completed cancer treatment. EMBody was co-created with young cancer survivors, paediatric oncologists with decades of clinical experience, and documentary filmmakers.

EMBody comprises three modules which include seven short films and accompanying reflection activities. The films feature young cancer survivors sharing their challenges of life after cancer and how their mindsets have supported them through these challenges. The films also feature oncology clinicians sharing their experience of the importance of mindsets in life after cancer, and psychological scientists who share information about what mindsets are and how they can be harnessed.

The main objective of the study is to assess whether a digital body mindset intervention (EMBody) can instil adaptive mindsets and improve health and wellbeing in young cancer survivors aged 16-25 years.

Researchers will compare the EMBody digital intervention with a waitlist attention control group to see if EMBody can instil adaptive mindsets and improve indicators of health and wellbeing in comparison to being enrolled in a study and completing study measures alone.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16-25 years
* Previously received a cancer diagnosis including but not limited to leukemia, Hodgkins/non-Hodgkins lymphoma, osteosarcoma, Ewing sarcoma, or CNS tumour
* Completed active, primary cancer treatment
* Are up to seven years off treatment

Exclusion Criteria:

* Significant cognitive impairment that would interfere with engagement with digital materials
* Not able read or write in English
* Active suicidal intent
* Currently receiving active treatment for primary or secondary cancer
* Completed cancer treatment more than seven years ago

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  The Young Adult Pediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL) measure assesses four domains of HRQOL using 23 items across separate subscales of physical, social, emotional and school functioning. For all items, individuals respond on a 5-point likert scale with an amended 7 day recall period (0= never a problem, 4= almost always a problem). Higher PedsQL 4.0 scores indicate better HRQOL.

SECONDARY OUTCOMES:
Body Mindsets | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  The Body Mindset Inventory (BMI-2) contains items that assess different mindsets about the body, capturing both adaptive and maladaptive mindsets. For all items, individuals respond on a 6-point Likert scale (6= strongly agree, 1= strongly disagree). Higher mean scores on each mindset subscale indicate greater endorsement of that mindset.
Illness Mindsets | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  The Illness Mindset Inventory (IMI) contains 9 items that assess different mindsets about the body and about cancer, capturing both adaptive ('manageable', 'opportunity') and maladaptive ('catastrophe') mindsets. For all items, individuals respond on a 6-point Likert scale (6= strongly agree, 1= strongly disagree). Higher mean scores on each mindset subscale indicate greater endorsement of that mindset.
The Functionality Appreciation Scale | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  The Functionality Appreciation Scale (FAS) (Alleva et al, 2017) contains 7-items that capture the overall appreciation of the body's ability to function to the extent that it can. Individuals respond to items on a 5-point Likert scale (1=strongly disagree, to 5=strongly agree). A total score is created by summing items where higher scores reflect a higher appreciation for the functionality of the body.
Pain | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  Items from the The Graded Chronic Pain Scale-Revised (Von Korff et al., 2020) and the body map from the Brief Pain Inventory (Cleeland et al, 1994) will be used to assess pain, including pain interference.
Hospital Anxiety and Depression Scale | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  The Hospital Anxiety and Depression Scale (HADS) contains 14-items assessing anxiety and depression symptoms with two separate subscales, each consisting of seven items. Items are rated from 0 to 3 and subscale scores range from 0 (no distress) to 21 (maximum distress).
Fear of Cancer Recurrence Inventory Short Form (FCRI-SF) | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  The Fear of Cancer Recurrence Inventory Short Form (FCRI-SF) contains 9-items assessing presence, frequency, intensity, and duration of fear of cancer recurrence thoughts and individual perceived risk of cancer recurrence. Items are rated on a 5-point likert scale and are amended to a 7 day recall period (0= not at all, 4= a great deal). Item five is reverse scored and total scores range from 0 to 36; higher scores reflect greater fear of cancer recurrence.
Post-Traumatic Growth Inventory (PTGI) | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  The Post-Traumatic Growth Inventory contains 21-items that evaluates positive changes after experiencing a stressful event such as cancer. Individuals respond on a 6-point Likert scale (0= I have not experienced this change as a result of my cancer experience - 6= I have experienced this change to a very great degree as a result of my cancer experience). A total score is created by summing all items. The scale also contains five factors and therefore separate scores can be created for each of these factors (relating to others, new possibilities, personal strength, spiritual change, appreciation of life).
Bodily Threat Monitoring Scale (BTMS) | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  The Bodily Threat Monitoring Scale (Heathcote et al, 2023) captures tendencies to monitor and appraise bodily sensations as symptomatic of something being wrong with one's body. The original scale includes 19-items, however a Short Form was used for this study. Each item is rated on a 5-point Likert scale (0= not at all like me, 4= entirely like me). Scores from items are summed and higher scores represent greater bodily threat monitoring.
Physical Activity | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  Physical activity will be captured using the Godin Leisure-Time Exercise Questionnaire (GLTEQ), which assesses physical activity throughout an individual's week based on four levels of activity intensity: strenuous, moderate, mild and sedentary. Higher scores indicate higher leisure-time physical activity.
The PedsQL Multidimensional Fatigue Scale in young adults | Assessed at all timepoints through study completion (2, 4, 6, 10, 18 weeks post-randomisation) and at the additional 12-month follow-up
  The PedsQL multidimensional fatigue scale captures general fatigue, sleep/rest fatigue and cognitive fatigue. This study uses the General Fatigue subscale. Respondents rate each of the 6 items on the General subscale a 5-point Likert scale ranging from 0 (never a problem) to 4 (almost always a problem). Scores are summed and higher scores indicate greater general levels of fatigue.
Global Impression of Change | Week 6 (T3)
  The Global Impression of Change (GIC) contains one item will be used to evaluate a patient's overall perception of improvement or deterioration over time from taking part in the EMBody study.

OTHER OUTCOMES:
Acceptability | Week 6 (T3).
  Nine items adapted from the Net Promoter Scale will capture acceptability of the EMBody intervention. Two additional open ended questions will also enable participants to provide written feedback on the intervention.
Adverse Events | Adverse Events Questions - T3 (week 6). Open Text Form - available freely to participants. PHQ9 - T0-T4 (baseline to week 10).
  Wileman et al 2024's adverse events and risk assessment protocol for digital trials has been amended to capture adverse events. Questions designed to capture adverse events (physical, psychological or otherwise) and suicidal ideation intent will be asked based on Wileman's 2024 protocol using the PHQ9 and an additional question asking about plan for those reporting intent. Participants will also have access to an open field text response prompting them to share any details of possible side effects or events related to their duration of taking part in the study. This will be accessible to participants 24/7 to capture further information about possible adverse events.
Heart Rate Variability | Assessed at baseline (T0), week 6 (T3), week 10 (T4), week 18 (T5).
  The HRV4Training app (www.hrv4training.com) will be used to capture 1 minute measurements of heart rate variability (HRV) using a mobile device camera while seated.
Healthcare Usage | Week 6 (T3).
  The UK Cancer Costs Questionnaire assess the financial impact of cancer on patients and their families. Costs from usage across services can be summed to indicate financial burden and cost associated with healthcare usage. Three additional items will be provided at T3 to the intervention group to capture whether participants have sought psychological support since receiving the intervention.
Storytelling | Week 6 (T3).
  Four items have been developed to capture the impact of intervention delivery through hearing stories from relatable others. Individuals respond on a 5-point likert scale from strongly disagree to strongly agree, and scores across items are summed to create a total score. Items will be provided for the intervention group only.
Qualtative Feedback | Week 6 (T3)
  Participants in the intervention arm will be invited to take part in an optional semi-structured interview to provide qualitative feedback on the EMBody intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C Heathcote, PhD, Principal Investigator — King's College London
Locations (1):
- The Royal Marsden, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with other researchers to comply with open science practices.
Time Frame: De-identified IPD will be shared on an online, open science data repository platform from the time that the study has been published and will be available indefinitely.
Access Criteria: De-identified IPD will be available open access.